CLINICAL TRIAL: NCT06066125
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of AK111 in the Treatment of Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of AK111 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-301
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Psoriasis; Skin Diseases
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK111 regimen 1 (Experimental)
  Interventions: Drug: AK111
- AK111 regimen 2 (Experimental)
  Interventions: Drug: AK111
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK111 — AK111 regimen 1- subcutaneous injection at week 0,1,2, 3,4 and every 4 weeks thereafter until week 48. The primary endpoint will be evaluated at week 12 and followed up to week 56.
  Arms: AK111 regimen 1
Drug: AK111 — AK111 regimen 2- subcutaneous injection at week 0,1,2, 3,4 and every 4 weeks thereafter until week 48. The primary endpoint will be evaluated at week 12 and followed up to week 56.
  Arms: AK111 regimen 2
Drug: Placebo — Placebo- subcutaneous injection at week 0,1,2, 3, 4 and week 8. AK111 regimen 2-subcutaneous injection every 4 weeks from week 12 to week 48. The primary endpoint will be evaluated at week 12 and followed up to week 56.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter phase III clinical study to evaluate the efficacy and safety of AK111 in the treatment of subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter phase III clinical study to evaluate the efficacy and safety of AK111 in the treatment of subjects with moderate to severe plaque psoriasis. Subjects will be randomized to receive AK111 or placebo subcutaneously and followed up to week 56.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years old.
2. Subjects diagnosed with moderate to severe plaque psoriasis with or without psoriatic arthritis.
3. At screening and baseline, PASI score ≥ 12 , Body Surface Area(BSA) ≥ 10%, sPGA ≥ 3.
4. Suitable for systematic therapy assessed by investigators.
5. Subjects who are women of childbearing potential must have a negative pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control during the study and for at least 6 months after the last study drug administration.

Exclusion Criteria:

1. Types of psoriasis other than chronic plaque-type psoriasis.
2. Drug-induced psoriasis.
3. Evidence of active TB. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment had initiated and maintained according to protocol.
4. Positive results of confirmatory test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or syphilis.
5. History of repeated chronic infection, had any serious infection or systemic infection within 2 months before screening.
6. Progressive or uncontrolled symptoms or signs of circulatory, respiratory, digestive, neuropsychiatric or psychological, hematological, endocrine and other systems before randomization.
7. History of malignant tumour within 5 years before screening.
8. Previous or current autoimmune diseases.
9. Allergic to any component of the investigational drug, or have had severe allergic reactions to monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who achieved at least 75% reduction in psoriasis area and severity index(PASI) score from baseline (PASI 75) and the percentage of subjects who achieved static physician global assessment(sPGA) 0/1 at week 12. | at week 12
  PASI is a combined assessment of a lesion severity and affected area into a single score: 0 (no disease) to 72(maximal disease). The body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for a final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%),and severity is estimated by clinical signs, erythema, induration and desquamation: scale 0 (none) to 4 (maximum).Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2, body: 0.3,legs: 0.4).PASI 50, PASI75 and PASI 90 were defined as participants achieving >= 50%, >= 75% or >= 90% improvement from baseline, respectively.The sPGA is an instrument providing a subjective evaluation of the overall severity of psoriasis, based on severity of induration, scaling, and erythema. The scores are: 0 = clear; 1 = minimal; 2 = mild; 3 = moderate; 4 = marked; 5 =severe.

SECONDARY OUTCOMES:
The percentage of subjects who achieved at least 90% reduction in PASI score from baseline (PASI 90) at week 12. | at week 12
The percentage of subjects who achieved PASI 75 and the percentage of subjects who achieved sPGA 0/1 at week 52. | at week 52

CONTACTS AND LOCATIONS:
Locations (34):
- China (34):
  - The first affiliated hospital of Bengbu Medical College, Bengbu, Anhui
  - The first affiliated hospital of wannan medical college, Wannan, Anhui
  - Affiliated hospital of Chongqing Three Gorges Medical College, Chongqing, Chongqing Municipality
  - Chongqing traditional Chinese medicine hospital (Daomenkou branch), Chongqing, Chongqing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen People's hospital, Shenzhen, Guangdong
  - The first affiliated hospital of Hainan Medical university, Haikou, Hainan
  - Nanyang First People's hospital national third class a hospital, Nanyang, Henan
  - Renmin hospital of Wuhan University Hubei general hospital, Wuhan, Hubei
  - Yichang central People's hospital, Yichang, Hubei
  - The third Xiangya hospital of Central South University, Changsha, Hunan
  - The frist People's hospital of Lianyungang, Lianyungang, Jiangsu
  - Dermatology Hospital of China Union Medical University, Nanjing, Jiangsu
  - The affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yancheng No.1 People's hospital, Yancheng, Jiangsu
  - Dermatology hospital of Jiangxi province, Nanchang, Jiangxi
  - The second hospital of Dalian Medical University, Dalian, Liaoning
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu hospital of the Fourth Military Medical University, Tanggu, Shanxi
  - West China school of medicine, West China hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin academy of traditional Chinese medicine affiliated hospita, Tianjin, Tianjin Municipality
  - Tianjin Medical University general hospital, Tianjin, Tianjin Municipality
  - Hangzhou first People's hospital, Hangzhou, Zhejiang
  - The first hospital of Jiaxing, Jiaxing, Zhejiang
  - Ningbo Huamei hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - The first affiliated hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing friendship hospital, Capital Medical University, Beijing
  - Peking University third hospital, Beijing
  - Guangdong provincial people's hospital, Guangdong
  - Affiliated hospital of Chengde Medical University, Hebei
  - The second affiliated hospital of Harbin Medical University, Heilongjiang
  - Xiangya hospital Central South University, Hunan
  - Huashan hospital, Fudan University, Shanghai
  - Shanghai skin disease hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No